CLINICAL TRIAL: NCT03699826
Title: Experimental Tinnitus Treatment With Transcranial Magnetic Stimulation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding source
Sponsor: Aaron Boes (Other)
Responsible Party: Sponsor-Investigator, Aaron Boes, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201808852
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Tinnitus
Keywords: transcranial magnetic stimulation; neuromodulation
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active TMS (Experimental): Active TMS stimulation administered for tinnitus symptoms (no sham stimulation).
  Interventions: Device: TMS for tinnitus

INTERVENTIONS:
Device: TMS for tinnitus — Targeted stimulation to decrease tinnitus symptom severity.

SUMMARY:
There are numerous conditions that may benefit from TMS but they lack definitive data from clinical trials with sufficient scientific rigor, which includes large, multi-site, randomized sham-controlled trials. This is the status for a variety of psychiatric and neurological disorders such as tinnitus, central pain, movement disorders, stroke rehabilitation, obsessive compulsive disorders, anxiety, schizophrenia, and addiction. In certain instances there may be sufficient evidence supporting the treatment efficacy of TMS that it is reasonable to offer TMS as an off-label treatment, a term for clinical treatments that have not received FDA approval but may nonetheless be helpful for patients. In other cases there is such a paucity of clinical trial data that the use of therapeutic TMS is less appropriate as a clinical treatment that the patient is charged for out of pocket and may cost several thousand dollars, but is better suited for clinically-oriented research. This has the added benefit of potentially helping the patient and providing investigators with additional information from which to inform future clinical trials. In this study the investigators propose to use TMS to treat tinnitus, for which few other treatments currently exist. Tinnitus affects approximately 1% of the population and can be debilitating for patients. Recent studies have shown some promise in reducing symptoms through neuromodulation, but results are variable and more research is needed to improve treatment protocols. The investigators plan to contribute to this body of research by taking an evidence-based approach to test whether TMS is effective at reducing symptoms of tinnitus. Each subject's MRI will be used to perform neuronavigated TMS stimulations while documenting changes in symptom severity with self-report questionnaires and symptom severity scales. If it is determined that a stimulation protocol is effective, 1-2 weeks of daily treatments will be scheduled as part of that subject's personalized treatment plan.

DETAILED DESCRIPTION:
1. Consent patients that have been referred to the Noninvasive Brain Stimulation Clinic at the University of Iowa.
2. Patients will complete the following before any treatments occur: Tinnitus Intake Questionnaire, Tinnitus Functional Index, Tinnitus Questionnaires, Iowa Tinnitus Primary Function, Clinical Global Improvement Scale.
3. Patients may undergo audiological assessment if they have not already been tested prior to the study.
4. Patients will be required to obtain an MRI prior to treatment to aid in neuronavigated stimulation unless there is have access to a previous clinical MRI for this purpose.
5. MRI images will be loaded into BrainSight or Localite, which are both frameless stereotactic systems for MRI-guided TMS localization. If no MRI is acquired, the subject's head will be transformed to MNI standard space within the software. Neuronavigation allows us to place specific stimulation targets onto each subjects's MRI. For this study, the investigators will be targeting left dorsolateral prefrontal cortex, auditory cortices, and auditory association cortices; all targets are placed anatomically by a neurologist. Infrared trackers on the subject's head and TMS coil allow for neuronavigated stimulation of anatomical targets on the cortex with millimeter precision.
6. The motor threshold of the subject will be assessed, which is the intensity of TMS required to elicit motor evoked potentials from the hand 50% of the time.
7. Subjects will be fitted with an EEG cap to record neural activity before, during, and after the initial test session.
8. Single TMS pulses or brief trains of repetitive TMS lasting a few seconds will be administered at 80 - 120% of motor threshold to targeted regions of the cerebral cortex and cerebellum. A typical experiment will last 30 minutes to 2 hours. The patients are told they can stop the experiment at any time.
9. After each stimulation, patients will be asked to rate any changes in symptom severity and whether any side effects were experienced (Tinnitus Questionnaires, Clinical Global Improvement Scale).
10. After the treatment session, the TMS pulse locations will be related to changes in symptom severity as measured by self-report. If any stimulation treatments were successful in reducing symptom severity, a treatment plan for that target will be discussed and follow-up treatments may be scheduled.
11. Follow up treatments will vary between patients but will typically consist of daily treatments for up to 4 weeks or until treatment response is sustained. The patient can withdraw from follow treatments at any time. Patients will be asked to complete the following at these visits: Tinnitus Functional Index, Tinnitus Questionnaires, Iowa Tinnitus Primary Function, Clinical Global Improvement Scale.

ELIGIBILITY:
Inclusion Criteria:

* tinnitus diagnosis

Exclusion Criteria:

* have epilepsy or a family history of epilepsy
* have implanted metal in or near their head
* have any history of brain injury or stroke
* have a tinnitus handicap inventory score of <38 (less than moderate handicap)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron D Boes, MD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS for Tinnitus: TMS for tinnitus: Open label study of neuro-navigated transcranial magnetic stimulation evaluating different stimulation sites and different stimulation protocols to decrease tinnitus symptom severity. Our goal was to evaluate whether a trial-and-error targeting session could be useful in selecting the stimulation site and frequency of stimulation before conducting daily treatments.
Period: Overall Study
Arm/Group | TMS for Tinnitus
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TMS for Tinnitus
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 65 [65 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement
Description: Clinical Global Improvement Scale (0-7 scale where 0=not assessed, 1=Very much improved, and 7= Very much worse
Time Frame: End of treatment course - 5 days
Population: single patient
Measure: Number; unit: score on a scale
Groups:
- TMS Treatment (Open Label, N = 1): TMS for tinnitus: Targeted stimulation to decrease tinnitus symptom severity.
Arm/Group | TMS Treatment (Open Label, N = 1)
Number analyzed (Participants) | 1
score on a scale | 4

ADVERSE EVENTS:
Time Frame: Adverse event data collected during TMS treatment course over a 1 week period.
Groups:
- TMS Treatment Arm: Open label study in single participant.
Arm/Group | TMS Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT03699826/Prot_001.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03699826/ICF_002.pdf